CLINICAL TRIAL: NCT01718951
Title: Golimumab Versus Pamidronate for the Treatment of Axial Spondyloarthropathy: a 48-week Randomized Controlled Trial
Brief Title: Golimumab Versus Pamidronate for the Treatment of Axial Spondyloarthropathy: a 48-week Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Chi Chiu Mok, Consultant, Tuen Mun Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREC/769/09
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Spondyloarthropathy
Keywords: spondyloarthropathy; ankylosing spondylitis
MeSH Terms: conditions — Spondylarthropathies; Spondylitis, Ankylosing | interventions — golimumab; Pamidronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- golimumab (Active Comparator): golimumab 50mg subcutaneous every 4 weeks
  Interventions: Drug: golimumab
- pamidronate (Active Comparator): Pamidronate (60mg) intravenously every 4 weeks
  Interventions: Drug: Pamidronate

INTERVENTIONS:
Drug: golimumab — golimumab
  Other Names: Simponi
  Arms: golimumab
Drug: Pamidronate — pamidronate
  Other Names: Aridia
  Arms: pamidronate

SUMMARY:
To compare the efficacy of golimumab with pamidronate in the treatment of axial spondyloarthropathy

DETAILED DESCRIPTION:
To compare the efficacy of golimumab with pamidronate in the treatment of non-radiological axial spondyloarthropathy

ELIGIBILITY:
Inclusion Criteria:

1. Subjects greater than 18 years of age
2. Fulfilling the latest classification criteria for axial spondyloarthropathy
3. Active spondylitis as defined by a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score of more than 4 despite treatment with non-steroid anti-inflammatory drugs for more than 3 months

Exclusion Criteria:

1. Major surgery (including joint surgery) within 8 weeks prior to study entry
2. History of treatment with anti-tumor necrosis factor agents or any investigational therapies within 12 months of study entry
3. Immunization with a live/attenuated vaccine within 4 weeks prior to study entry
4. Active current bacterial, viral, fungal, mycobacterial or other infections at study entry
5. Chronic hepatitis B or hepatitis C carriers
6. History of malignancies, including solid tumors and hemic malignancies
7. History of congestive heart failure
8. History of demyelinating disorders
9. History of peripheral neuropathy
10. Pregnant women or lactating mothers
11. Baseline liver parenchymal enzymes elevated to more than 2 times normal
12. Absolute lymphocyte count less than 500/mm3
13. Serum creatinine level of more than 200umol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-08; Primary Completion 2014-03 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Assessment of SpondyloArthritis international Society criteria (ASAS)-20 response response | week 48
  Proportion of patients who achieve the Assessment of SpondyloArthritis international Society criteria (ASAS)-20 response

SECONDARY OUTCOMES:
Changes in MRI spinal inflammation scores | week 24 and 48
  Changes in MRI spinal inflammation scores

CONTACTS AND LOCATIONS:
Locations (1):
- Tuen Mun Hospital, Hong Kong, Hong Kong